CLINICAL TRIAL: NCT01581983
Title: Mindfulness Meditation Format Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Helane Wahbeh, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00008355
Record Dates: First submitted 2012-04-07; First posted 2012-04-20 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Posttraumatic Stress Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Internet Mindfulness Meditation (Experimental)
  Interventions: Behavioral: Internet Mindfulness Meditation
- Individual Mindfulness Meditation (Experimental)
  Interventions: Behavioral: Individual Mindfulness Meditation

INTERVENTIONS:
Behavioral: Internet Mindfulness Meditation — one hour session each week for six weeks
  Arms: Internet Mindfulness Meditation
Behavioral: Individual Mindfulness Meditation — one hour session each week for six weeks
  Arms: Individual Mindfulness Meditation

SUMMARY:
The purpose of this study is to assess feasibility of an internet and individual format of mindfulness meditation in people with posttraumatic stress disorder (PTSD) and depression symptoms

DETAILED DESCRIPTION:
Internet and individual formats of mindfulness meditation have not been previously evaluated. In order establish feasibility of such formats a pilot study is need. The current study will randomize up to 20 people with PTSD and depression symptoms and evaluate changes in PTSD and depression symptoms from before to after the internet and individual mindfulness meditation interventions.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Age 25-65
* Access to internet
* PTSD symptoms (score >14 on PTSD screen)
* Depression symptoms (endorsement of one question on depression screen)
* Stable on medications six weeks prior to the study
* Willing to be stable on medications during study

Exclusion Criteria:

* Significant potentially life-limiting acute medical illness
* Risk for suicide
* >2 drinks/day of alcohol and street drug use besides marijuana
* Current daily meditation practice

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist | Change from baseline to week 7.
  The Posttraumatic Stress Disorder Checklist will be administered immediately before their first intervention session and within one week of their last intervention session. The primary outcome is the change in score on this instrument from baseline to week 7.
Beck Depression Inventory | Change from Baseline to Week 7
  The Beck Depression Inventory will be administered immediately before their first intervention session and within one week of their last intervention session. The primary outcome is the change in score on this instrument from baseline to week 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States